CLINICAL TRIAL: NCT05527327
Title: Pannus Retraction for Ultrasound Evaluation of the Obese Gravida: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1935904-1
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Pregnancy Complications; Fetal Anomaly; Pannus
Keywords: obesity; pregnancy; pannus; ultrasound; fetal anomaly
MeSH Terms: conditions — Obesity; Pregnancy Complications; Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: All prospective participants will receive the intervention for one occurrence. Retrospective participants' results will be observed without any intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective arm (Experimental): All prospective participants will be consented to use of the intervention, a pannus retractor at time of detailed obstetric ultrasound.
  Interventions: Device: traxi® Panniculus Retractor

INTERVENTIONS:
Device: traxi® Panniculus Retractor — This is an adhesive medical device designed to retract a pannus during cesarean section. It will be applied to prospective participants according to manufacturer instructions, just prior to the detailed anatomic ultrasound.

SUMMARY:
Pregnancies complicated by obesity have an increased risk of multiple pregnancy complications, including structural fetal anomalies. Therefore, maternal obesity (BMI ≥30 kg/m2) is an indication for a detailed anatomic ultrasound examination. Ultrasound is a critical tool for the detection of congenital anomalies; however, obesity makes ultrasound examinations technically challenging.

The primary objective of this ambidirectional cohort pilot study is to evaluate whether utilization of a pannus retractor is associated with increased rates of detailed anatomic ultrasound completion amongst pregnant patients with a body mass index (BMI) greater than or equal to 40 kg/m2. Retrospective data will be collected for 100 patients with a BMI of 40 kg/m2 or greater to assess the baseline rate of completion of 16 components of the detailed anatomic survey prior to the intervention. We plan to enroll 20 patients into a prospective pilot to the intervention arm. The intervention is placement of an adhesive medical device, the traxi® Panniculus Retractor (Laborie, Portsmouth, New Hampshire), which was developed for pannus retraction during cesarean section. Adequacy of anatomic ultrasound completion will be based upon 16 pre-defined views from the anatomic survey. Ultrasound completion rates from the prospective cohort of participants that undergo ultrasound evaluation using a pannus retractor will be compared to a historical cohort without pannus retractor use. We hypothesize that use of a pannus retractor for pregnant participants with BMI greater than or equal to 40 kg/m2 increases the rate of anatomical ultrasound completion.

DETAILED DESCRIPTION:
Aim 1: Determine the completion rate of detailed obstetric ultrasound when using the pannus retractor device adhesive for participants with BMI of 40 kg/m2 or greater. Retrospective data will be collected for 100 patients with a BMI of 40 kg/m2 or greater to assess the baseline rate of completion of 16 components of the detailed anatomic survey. We will prospectively enroll twenty participants with BMI of at least 40 kg/m2 who consent to having a pannus retractor device adhesive placed for their anatomic ultrasound exam. Inclusion and exclusion criteria will be followed as detailed elsewhere. Participant measurements including current height, weight, and pannus grade will be recorded. The pannus retractor device adhesive will be placed by research personnel and sonographers who have been trained in proper application of the device, per manufacturer's instructions. The start time of adhesive application will be recorded. The ultrasound exam will then proceed as a routine ultrasound exam, except for two additional ultrasound measurements. Using no pressure, the distance from ultrasound probe to the amniotic cavity will be measured with and without the pannus retractor in place. Other collection variables will be available from chart review, namely age, race, ethnicity, insurance status, estimated due date, pre-pregnancy BMI, BMI at first obstetric visit, diabetic status, smoking status, parity, prior abdominal surgical status, date of ultrasound, fetal presentation, placental location, sonographer, reading physician, time of first and last ultrasound image acquisition, and whether transvaginal imaging was used. The outcome measure of interest, completion of adequate visualization of sixteen views, will be available from review of the final ultrasound report. The rate of completed studies from the prospective population will be compared to historical data to determine if Aim 1 hypothesis is true.

Aim 2: Determine changes to the sonographer experience for the 20 patients enrolled in the prospective cohort portion of this project. A survey will be administered to the sonographers who perform the ultrasounds with the pannus retractor adhesive in use. The amount of discomfort experienced in their arm or shoulder while scanning, their confidence in the quality of their images, and whether the ultrasound was made easier by use of the adhesive will be assessed by a Likert scale with space for free text comments.

Aim 3: Evaluate the participant experience for the 20 patients enrolled in the prospective cohort portion of this project. The comfort, satisfaction and enjoyment of the ultrasound experience will be assessed by a Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients presenting for detailed anatomic ultrasound with a BMI of at least 40 kg/m2
* English or Spanish speaking
* BMI of at least 40.0 kg/m2 at first obstetric visit during this pregnancy
* Gestational age between 18 weeks 0 days to 23 weeks 6 days

Exclusion Criteria:

* Patients who have already had an anatomy ultrasound during the same pregnancy with our department
* History of tape/adhesive allergy
* Multifetal gestation
* Known intrauterine fetal demise

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Complete ultrasound study (yes/no) | Up to one month from each individual's participation
  The ultrasound report will be evaluated to determine if the following elements were adequately visualized: lateral ventricles, cerebellum, cavum septum pellucidum, face, four chamber view, right outflow tract, left outflow tract, three vessel view, three vessel trachea view, spine, ventral wall, umbilical cord, stomach, left kidney, right kidney, bladder. If any one or more of these elements are not adequately visualized, the study will be interpreted as "incomplete." The proportion of complete to incomplete studies will be compared between the retrospective and prospective cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pasko, MD, Principal Investigator — Prisma Health Maternal-Fetal Medicine
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
All study investigators will have access to the database management system that includes IPD. Only de-identified results will be distributed after analysis.

REFERENCES:
- [Background] Lashen H, Fear K, Sturdee DW. Obesity is associated with increased risk of first trimester and recurrent miscarriage: matched case-control study. Hum Reprod. 2004 Jul;19(7):1644-6. doi: 10.1093/humrep/deh277. Epub 2004 May 13. PMID 15142995
- [Background] Stothard KJ, Tennant PW, Bell R, Rankin J. Maternal overweight and obesity and the risk of congenital anomalies: a systematic review and meta-analysis. JAMA. 2009 Feb 11;301(6):636-50. doi: 10.1001/jama.2009.113. PMID 19211471
- [Background] Racusin D, Stevens B, Campbell G, Aagaard KM. Obesity and the risk and detection of fetal malformations. Semin Perinatol. 2012 Jun;36(3):213-21. doi: 10.1053/j.semperi.2012.05.001. PMID 22713503
- [Background] AIUM Practice Parameter for the Performance of Detailed Second- and Third-Trimester Diagnostic Obstetric Ultrasound Examinations. J Ultrasound Med. 2019 Dec;38(12):3093-3100. doi: 10.1002/jum.15163. No abstract available. PMID 31736130
- [Background] Weichert J, Hartge DR. Obstetrical sonography in obese women: a review. J Clin Ultrasound. 2011 May;39(4):209-16. doi: 10.1002/jcu.20767. Epub 2010 Dec 7. PMID 21480286
- [Background] Dashe JS, McIntire DD, Twickler DM. Effect of maternal obesity on the ultrasound detection of anomalous fetuses. Obstet Gynecol. 2009 May;113(5):1001-1007. doi: 10.1097/AOG.0b013e3181a1d2f5. PMID 19384114
- [Background] Obesity in Pregnancy: ACOG Practice Bulletin, Number 230. Obstet Gynecol. 2021 Jun 1;137(6):e128-e144. doi: 10.1097/AOG.0000000000004395. PMID 34011890
- [Background] Dashe JS, McIntire DD, Twickler DM. Maternal obesity limits the ultrasound evaluation of fetal anatomy. J Ultrasound Med. 2009 Aug;28(8):1025-30. doi: 10.7863/jum.2009.28.8.1025. PMID 19643785
- [Background] Thornburg LL, Miles K, Ho M, Pressman EK. Fetal anatomic evaluation in the overweight and obese gravida. Ultrasound Obstet Gynecol. 2009 Jun;33(6):670-5. doi: 10.1002/uog.6401. PMID 19479682
- [Background] Pasko DN, Wood SL, Jenkins SM, Owen J, Harper LM. Completion and Sensitivity of the Second-Trimester Fetal Anatomic Survey in Obese Gravidas. J Ultrasound Med. 2016 Nov;35(11):2449-2457. doi: 10.7863/ultra.15.11057. Epub 2016 Oct 3. PMID 27698181
- [Background] Simmons PM, Wendel MP, Whittington JR, San Miguel K, Ounpraseuth ST, Magann EF. Accuracy and Completion Rate of the Fetal Anatomic Survey in the Super Obese Parturient. J Ultrasound Med. 2021 Oct;40(10):2047-2051. doi: 10.1002/jum.15582. Epub 2020 Dec 5. PMID 33277924